CLINICAL TRIAL: NCT02443688
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy, Safety, and Tolerability of CTX-4430 Administered Orally Once-Daily for 48 Weeks in Adult Patients With Cystic Fibrosis
Brief Title: EMPIRE CF: A Phase 2 Study to Evaluate the Efficacy, Safety, and Tolerability of CTX-4430 in Adult Cystic Fibrosis (CF) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celtaxsys, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTX-4430-CF-201
Record Dates: First submitted 2015-05-08; First posted 2015-05-14 (Estimated); Results first posted 2019-07-25 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — acebilustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 50 mg CTX-4430 (Experimental): Once daily oral capsule for 48 weeks
  Interventions: Drug: CTX-4430
- 100 mg CTX-4430 (Experimental): Once daily oral capsule for 48 weeks
  Interventions: Drug: CTX-4430
- Matching Placebo (Placebo Comparator): Once daily oral capsule for 48 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CTX-4430
  Arms: 100 mg CTX-4430; 50 mg CTX-4430
Drug: Placebo
  Arms: Matching Placebo

SUMMARY:
This study is a Phase 2, double-blind, randomized, placebo-controlled study to evaluate the safety and efficacy of CTX-4430 administered once-daily for 48 weeks for treatment of CF.

DETAILED DESCRIPTION:
This study is a Phase 2, double-blind, randomized, placebo-controlled study to evaluate the safety and efficacy of CTX-4430 administered once-daily for 48 weeks for treatment of CF. A total of 195 pulmonary CF patients that meet all the inclusion and no exclusion criteria and provide written informed consent will be randomized to receive 50 mg CTX-4430, 100 mg CTX-4430, or placebo in a 1:1:1 ratio. Follow-up visits will be conducted approximately every 4 weeks from Week 4 to Week 52 (4 weeks after completion of treatment).

ELIGIBILITY:
Inclusion Criteria:

* Forced expiratory volume at one second (FEV1) ≥50 percent predicted at Screening
* At least 1 pulmonary exacerbation in the 12 months before Screening

Exclusion Criteria:

* Pregnant or nursing women
* Medical condition that is unstable, could be adversely impacted by participation in the study, or could impact assessment of the study results
* History of organ transplantation
* History of alcoholism or drug abuse within 2 years before Screening
* Regular use of a high-dose NSAID within 60 days before Screening

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2015-10-30 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Rowe, MD, Principal Investigator — University of Alabama at Birmingham, USA; Stuart Elborn, MD, Principal Investigator — Royal Brompton Hospital, London UK
Locations (75):
- United States (39):
  - University of Alabama, Birmingham, Alabama
  - Providence Health and Services, Anchorage, Alaska
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Pediatric Pulmonary and Cystic Fibrosis Clinic, Stanford University, Palo Alto, California
  - University of California Davis Medical Center, Sacramento, California
  - National Jewish Health, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Central Florida Pulmonary Group, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - St. Francis Medical Center, Peoria, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Maine Medical Center, Portland, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Harper University Hospital, Detroit, Michigan
  - Spectrum Health Butterworth Campus, Grand Rapids, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of New Mexico, Albuquerque, New Mexico
  - Albany Medical College, Albany, New York
  - Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Wake Forest Hospital, Winston-Salem, North Carolina
  - UC Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health & Sciences University, Portland, Oregon
  - Hershey Medical Center, Hershey, Pennsylvania
  - Drexel University, Philadelphia, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Sanford Clinical Research, Sioux Falls, South Dakota
  - Universiy of Tennessee Medical Center UHS, Knoxville, Tennessee
  - Dell Children's Medical Center, Austin, Texas
  - Cook Children's Hospital, Fort Worth, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (2):
  - Hôpital Erasme, Brussels
  - UZ Leuven, Leuven
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - Ottawa Hospital, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
- France (5):
  - Centre hospitalier de Dunkerque, Dunkirk
  - Hôpital Albert Michallon, Grenoble
  - Hopital Arnaud de Villeneuve, Montpellier
  - Hôpital Cochin, Paris
  - CH Lyon Sud, Pierre-Bénite
- Germany (10):
  - Charite' University, Berlin
  - Krankenhaus Donaustauf, Donaustauf
  - Carl-Gustav-Klinikum Dresden, Mukoviszidose Centrum "Christiane Herzog", Dresden
  - Ruhrlandklinik Essen, Essen
  - Institut für klinische Forschung Pneumologie, Frankfurt
  - Klinikum der Johann Wolfgang Goethe-Universität, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Jena CF Centre, Jena
  - Lungenärztliche Praxis München-Pasing, München-Pasing
  - Klinikum Stuttgart CF Ambulanz, Stuttgart
- Italy (5):
  - Ospedali Riuniti di Ancona, Ancona
  - Azienda Ospedaliero Universitaria, Catania
  - Azienda Ospedaliera A Meyer, Florence
  - IRCCS Ospedale Pediatrico Bambino, Rome
  - Ospedale Civile Maggiore, Verona
- United Kingdom (11):
  - Belfast City Hospital, Belfast
  - Bristol Royal Infirmary, Bristol
  - Llandough Hospital, Cardiff
  - St James's University Hospital, Leeds
  - Liverpool Heart and Chest Hospital, Liverpool
  - King's College Hospital, London
  - Royal Brompton Hospital, London
  - University Hospital of South Manchester, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - University Hospital Southampton, Southampton
  - Royal Stoke University Hospital, Stoke-on-Trent

RESULTS

PARTICIPANT FLOW:
Groups:
- 100 mg CTX-4430; 50 mg CTX-4430: Once daily oral capsule for 48 weeks
  CTX-4430
- Matching Placebo: Once daily oral capsule for 48 weeks
  Placebo
Period: Overall Study
Arm/Group | 100 mg CTX-4430 | 50 mg CTX-4430 | Matching Placebo
Started | 66 | 67 | 67
Completed | 54 | 58 | 55
Not Completed | 12 | 9 | 12
Not completed — Adverse Event | 2 | 3 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Physician Decision | 3 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 3 | 4
Not completed — Non-compliance with study drug | 1 | 2 | 4
Not completed — Sponsor Request | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: One subject in the matching placebo cohort was randomized but did not take any study drug. Therefore, the matching placebo group has 66 subjects listed instead of 67 subjects making it a total of 199 subjects who received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 100 mg CTX-4430 | 50 mg CTX-4430 | Matching Placebo | Total
Number analyzed (Participants) | 66 | 67 | 66 | 199
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 6 | 4 | 12
  Between 18 and 65 years | 64 | 61 | 62 | 187
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (3.24) | 23.7 (3.64) | 23.2 (3.38) | 23.7 (3.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 38 | 33 | 101
  Male | 36 | 29 | 33 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 0 | 7
  Not Hispanic or Latino | 61 | 65 | 66 | 192
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 0 | 4
  White | 62 | 62 | 66 | 190
  More than one race | 3 | 2 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
On cystic fibrosis transmembrane conductance regulator (CFTR) Modulator Therapy: Yes [Count of Participants; unit: Participants] | 21 | 22 | 19 | 62
On CFTR Modulator Therapy: No [Count of Participants; unit: Participants] | 45 | 45 | 47 | 137
Number of Pulmonary Exacerbations in the year prior to Screening [Mean (Standard Deviation); unit: pulmonary Exacerbations/year] | 2.32 (1.947) | 2.13 (1.466) | 1.94 (1.357) | 2.13 (1.609)

OUTCOME MEASURES:

1. Primary Outcome: Difference From Placebo in Absolute Change From Baseline in Forced Expiratory Volume in 1 Second Percent Predicted (ppFEV1)
Description: Difference from Placebo in absolute change from Baseline at Week 48 was assessed for FEV1 percent predicted.
Time Frame: Baseline, Week 48
Population: Full Analysis Population - All subjects randomized to and receiving at least 1 dose of assigned treatment. The primary analysis was based upon the pooled results of the 100mg and 50mg doses.
Measure: Mean (95% Confidence Interval); unit: FEV1 percent predicted
Groups:
- Pooled CTX-4430: The average of the Week 48 absolute change from Baseline in FEV1 percent predicted for the two CTX-4430 doses.
Arm/Group | 100 mg CTX-4430 | 50 mg CTX-4430 | Pooled CTX-4430 | Matching Placebo
Number analyzed (Participants) | 66 | 67 | 133 | 66
FEV1 percent predicted | -1.30 [-3.22 to 0.62] | -3.76 [-5.65 to -1.86] | -2.53 [-3.88 to -1.18] | -2.69 [-4.63 to -0.75]
Statistical Analysis 1: Comparison: 100 mg CTX-4430; Test type: Other — Single Group Difference from Placebo Mean Change from Baseline with 95% confidence interval (CI); ANOVA; Mean Difference (Final Values) = 1.39, 95% CI 2-sided [-1.34 to 4.12], Standard Error of Mean 1.38
Statistical Analysis 2: Comparison: 50 mg CTX-4430; Test type: Other — Single Group Difference from Placebo Mean Change from Baseline with 95% CI; ANOVA; Mean Difference (Final Values) = -1.07, 95% CI 2-sided [-3.78 to 1.64], Standard Error of Mean 1.37
Statistical Analysis 3: Comparison: Pooled CTX-4430; Test type: Superiority — Difference from placebo of pooled arms (100mg CTX-4430 and 50mg CTX-4430) in change from baseline in ppFEV1 at Week 48; p = 0.45, ANOVA — 0.1 alpha level (2-sided) prespecified; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-2.20 to 2.50], Standard Error of Mean 1.2

2. Secondary Outcome: Number of Pulmonary Exacerbations Through 48 Weeks
Description: Rate of protocol-defined pulmonary exacerbations reported through the Week 48/Early Termination visit will be annualized where a year is defined by 52 weeks and will be analyzed using a negative binomial regression.
Time Frame: Week 48
Population: Full Analysis Population - All subjects randomized to and receiving at least 1 dose of assigned treatment. The statistical analysis plans states the two active doses will be compared to placebo individually as well as pooled.
Measure: Mean (95% Confidence Interval); unit: pulmonary exacerbations per year
Groups:
- Pooled CTX-4430: Once daily oral 100mg and 50mg pooled results
Arm/Group | 100 mg CTX-4430 | 50 mg CTX-4430 | Pooled CTX-4430 | Matching Placebo
Number analyzed (Participants) | 66 | 67 | 133 | 66
pulmonary exacerbations per year | 1.57 [1.22 to 2.02] | 1.46 [1.13 to 1.89] | 1.51 [1.26 to 1.81] | 1.56 [1.21 to 2.01]
Statistical Analysis 1: Comparison: 100 mg CTX-4430; Test type: Other — Single Group Rate with 95% CI; see Estimation Comment below = 1.57, 95% CI 2-sided [1.22 to 2.02], Standard Error of Mean 0.20 — Estimated using negative binomial distribution by treatment group unadjusted for multiple comparisons
Statistical Analysis 2: Comparison: 50 mg CTX-4430; Test type: Other — Single Group Rate with 95% CI; see Estimation Comment below = 1.46, 95% CI 2-sided [1.13 to 1.89], Standard Error of Mean 0.19 — Estimated using negative binomial distribution by treatment group unadjusted for multiple comparisons
Statistical Analysis 3: Comparison: Matching Placebo; Test type: Other — Single Group Rate with 95% CI; see Estimation Comment below = 1.56, 95% CI 2-sided [1.21 to 2.01], Standard Error of Mean 0.20 — Estimated using negative binomial distribution by treatment group unadjusted for multiple comparisons
Statistical Analysis 4: Comparison: Pooled CTX-4430; Test type: Other — Pooled Group Rate with 95% CI; see Estimation Comment below = 1.51, 95% CI 2-sided [1.26 to 1.81], Standard Error of Mean 0.14 — Estimated using negative binomial distribution unadjusted for multiple comparisons

3. Secondary Outcome: Hazard Ratio Pulmonary Exacerbation While in the Study
Description: Hazard Ratio of pulmonary exacerbation versus placebo for all subjects. Pulmonary exacerbations are defined as treatment with oral, inhaled, or intravenous antibiotic(s) for ≥4 of symptoms/signs per the modified Fuchs criteria.
Time Frame: Week 48
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: hazard ratio
Arm/Group | 100 mg CTX-4430 | 50 mg CTX-4430 | Pooled CTX-4430
Number analyzed (Participants) | 66 | 67 | 133
hazard ratio | 0.88 [0.576 to 1.339] | 0.86 [0.563 to 1.308] | 0.87 [0.605 to 1.246]
Statistical Analysis 1: Comparison: 100 mg CTX-4430; Test type: Other — 95% 2-sided confidence interval for the Hazard Ratio relative to Placebo unadjusted for multiple comparisons; Regression, Cox; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.58 to 1.34], Standard Error of Mean 0.19
Statistical Analysis 2: Comparison: 50 mg CTX-4430; Test type: Other — 95% 2-sided confidence interval for the Hazard Ratio relative to Placebo unadjusted for multiple comparisons; Regression, Cox; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.56 to 1.31], Standard Error of Mean 0.18
Statistical Analysis 3: Comparison: 100 mg CTX-4430 vs 50 mg CTX-4430; Test type: Other — 95% 2-sided confidence interval for the Hazard Ratio Relative to Placebo unadjusted for multiple comparisons; Regression, Cox; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.61 to 1.25], Standard Error of Mean 0.16

4. Secondary Outcome: Subjects Without a Pulmonary Exacerbation While in the Study
Description: Subjects who did not experience a protocol-defined pulmonary exacerbation during the study
Time Frame: Week 48
Population: Full Analysis Population - All subjects randomized to and receiving at least 1 dose of assigned treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | 100 mg CTX-4430 | 50 mg CTX-4430 | Pooled CTX-4430 | Matching Placebo
Number analyzed (Participants) | 66 | 67 | 133 | 66
Participants | 25 | 26 | 51 | 20

5. Secondary Outcome: Relative Change (Percent Change) From Baseline in ppFEV1
Description: Percent change from Baseline for ppFEV1 at 48 weeks was assessed.
Time Frame: Baseline, Week 48
Population: Full Analysis Population - All subjects randomized to and receiving at least 1 dose of assigned treatment. (Observed Data). The statistical analysis plans states the two active doses will be compared to placebo individually as well as pooled.
Measure: Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | 100 mg CTX-4430 | 50 mg CTX-4430 | Pooled CTX-4430 | Matching Placebo
Number analyzed (Participants) | 59 | 59 | 118 | 57
percent change from baseline | -2.38 [-5.37 to 0.60] | -4.81 [-7.84 to -1.79] | -3.60 [-5.72 to -1.47] | -3.40 [-6.59 to -0.22]

6. Secondary Outcome: Change From Baseline at 48 Weeks for Forced Vital Capacity Percent Predicted (FVC) and FEF25-75% (Forced Expiratory Flow During the Middle Half of the Forced Vital Capacity) Percent Predicted
Time Frame: Baseline, Week 48
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: absolute change of percent predicted
Arm/Group | 100 mg CTX-4430 | 50 mg CTX-4430 | Pooled CTX-4430 | Matching Placebo
Number analyzed (Participants) | 59 | 59 | 118 | 57
absolute change of percent predicted
  Forced vital capacity (FVC) percent predicted | -1.57 [-3.37 to 0.23] | -2.06 [-3.88 to -0.25] | -1.82 [-3.10 to -0.54] | -1.41 [-3.32 to 0.51]
  Forced expiratory flow(FEF25-75%)percent predicted | -1.61 [-4.26 to 1.03] | -4.79 [-7.46 to -2.11] | -3.20 [-5.08 to -1.32] | -4.38 [-7.20 to -1.57]

7. Secondary Outcome: Change From Baseline for Specified Biomarkers
Description: Results were only calculated in subjects who had a verifiable result at the Baseline and Week 48 visits.
Time Frame: Baseline, Week 48
Population: Full Analysis Population - All subjects randomized to and receiving at least 1 dose of assigned treatment and who had results at Baseline and Week 48. The statistical analysis plans states the two active doses will be compared to placebo individually as well as pooled.
Measure: Mean (95% Confidence Interval); unit: log10(mcg/mL)
Arm/Group | 100 mg CTX-4430 | 50 mg CTX-4430 | Pooled CTX-4430 | Matching Placebo
Number analyzed (Participants) | 66 | 67 | 133 | 66
log10(mcg/mL)
  Sputum DNA: number analyzed (Participants) | 33 | 42 | 75 | 42
  Sputum DNA | 0.06 [-0.13 to 0.25] | 0.17 [0.01 to 0.34] | 0.12 [-0.01 to 0.24] | -0.05 [-0.22 to 0.12]
  Sputum Elastase: number analyzed (Participants) | 33 | 43 | 76 | 41
  Sputum Elastase | -0.02 [-0.20 to 0.16] | 0.17 [0.02 to 0.33] | 0.08 [-0.04 to 0.20] | -0.08 [-0.25 to 0.08]

8. Secondary Outcome: Change From Baseline for C-reactive Protein (Hs-CRP)
Description: Results were only calculated in subjects who had a verifiable result at the Baseline and Week 48 visits.
Time Frame: Baseline, Week 48
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | 100 mg CTX-4430 | 50 mg CTX-4430 | Pooled CTX-4430 | Matching Placebo
Number analyzed (Participants) | 51 | 55 | 106 | 51
mg/dL | 2.16 [-1.84 to 6.16] | -0.33 [-4.21 to 3.56] | 0.92 [-1.87 to 3.70] | -1.87 [-5.91 to 2.17]

9. Other Pre Specified Outcome: Number of Pulmonary Exacerbation Per Year for Participants With ppFEV1 >75 at Baseline
Description: as for outcome 2
Time Frame: Week 48
Population: Population of subjects with Baseline ppFEV1 >75. The statistical analysis plans states the two active doses will be compared to placebo individually as well as combined. The statistical analysis plans states the two active doses will be compared to placebo individually as well as pooled.
Measure: Mean (95% Confidence Interval); unit: pulmonary exacerbations per year
Arm/Group | 100 mg CTX-4430 | 50 mg CTX-4430 | Pooled CTX-4430 | Matching Placebo
Number analyzed (Participants) | 22 | 25 | 47 | 24
pulmonary exacerbations per year | 0.84 [0.49 to 1.44] | 1.28 [0.84 to 1.96] | 1.04 [0.74 to 1.46] | 1.61 [1.07 to 2.42]
Statistical Analysis 1: Comparison: 100 mg CTX-4430; Test type: Other — Single Group Rate with 95% CI; see Estimation Comment below = 0.84, 95% CI 2-sided [0.49 to 1.44], Standard Error of Mean 0.23 — Estimated using negative binomial distribution by treatment group unadjusted for multiple comparisons
Statistical Analysis 2: Comparison: 50 mg CTX-4430; Test type: Other — Single Group Rate with 95% CI; see Estimation Comment below = 1.28, 95% CI 2-sided [0.84 to 1.96], Standard Error of Mean 0.28 — Estimated using negative binomial distribution by treatment group unadjusted for multiple comparisons
Statistical Analysis 3: Comparison: Matching Placebo; Test type: Other — Single Group Rate with 95% CI; see Estimation Comment below = 1.61, 95% CI 2-sided [1.07 to 2.42], Standard Error of Mean 0.34 — Estimated using negative binomial distribution by treatment group unadjusted for multiple comparisons
Statistical Analysis 4: Comparison: Pooled CTX-4430; Test type: Other — Group Rate with 95% CI; see Estimation Comment below = 1.04, 95% CI 2-sided [0.74 to 1.46], Standard Error of Mean 0.18 — Estimated using negative binomial distribution by treatment group unadjusted for multiple comparisons

10. Other Pre Specified Outcome: Hazard Ratio Pulmonary Exacerbation for Participants With ppFEV1 >75 at Baseline
Description: Hazard ratio of pulmonary exacerbation versus placebo for all subjects
Time Frame: Week 48
Population: Population of subjects with Baseline ppFEV1 >75. The statistical analysis plan states the two active doses will be compared to placebo individually as well as pooled.
Measure: Number (95% Confidence Interval); unit: hazard ratio
Arm/Group | 100 mg CTX-4430 | 50 mg CTX-4430 | Pooled CTX-4430
Number analyzed (Participants) | 22 | 25 | 47
hazard ratio | 0.52 [0.245 to 1.101] | 0.62 [0.304 to 1.274] | 0.57 [0.307 to 1.051]
Statistical Analysis 1: Comparison: 100 mg CTX-4430; Test type: Other — 95% 2-sided confidence interval for the Hazard Ratio Relative to Placebo unadjusted for multiple comparisons; Regression, Cox; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.25 to 1.10], Standard Error of Mean 0.20
Statistical Analysis 2: Comparison: 50 mg CTX-4430; Test type: Other — 95% 2-sided confidence interval for the Hazard Ratio Relative to Placebo unadjusted for multiple comparisons; Regression, Cox; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.30 to 1.27], Standard Error of Mean 0.18
Statistical Analysis 3: Comparison: 100 mg CTX-4430 vs 50 mg CTX-4430; Test type: Other — 95% 2-sided confidence interval for the Hazard Ratio Relative to Placebo unadjusted for multiple comparisons; Regression, Cox; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.31 to 1.05], Standard Error of Mean 0.18

11. Other Pre Specified Outcome: Subjects Without a Pulmonary Exacerbation by Participants With ppFEV1 >75 at Baseline
Description: Subjects who did not experience a protocol-defined pulmonary exacerbation during the study.
Time Frame: Week 48
Population: Population of subjects with Baseline ppFEV1 >75.
Measure: Count of Participants; unit: Participants
Arm/Group | 100 mg CTX-4430 | 50 mg CTX-4430 | Pooled CTX-4430 | Matching Placebo
Number analyzed (Participants) | 22 | 25 | 47 | 24
Participants | 11 | 12 | 23 | 6

12. Other Pre Specified Outcome: Number of Pulmonary Exacerbation by Subjects if Taking CFTR-Modulator Therapy at Baseline
Description: as for outcome 2
Time Frame: Week 48
Population: Population of subjects taking CFTR modulating therapy at Baseline. The statistical analysis plans states the two active doses will be compared to placebo individually as well as pooled.
Measure: Mean (95% Confidence Interval); unit: pulmonary exacerbations per year
Arm/Group | 100 mg CTX-4430 | 50 mg CTX-4430 | Pooled CTX-4430 | Matching Placebo
Number analyzed (Participants) | 21 | 22 | 43 | 19
pulmonary exacerbations per year | 1.24 [0.78 to 1.96] | 1.08 [0.67 to 1.74] | 1.16 [0.83 to 1.61] | 1.45 [0.91 to 2.31]

13. Other Pre Specified Outcome: Hazard Ratio Pulmonary Exacerbation by Subjects if Taking CFTR-Modulator Therapy at Baseline
Description: Hazard Ratio pulmonary exacerbation versus placebo for all subjects taking CFTR-modulating therapy at Baseline
Time Frame: Week 48
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: hazard ratio
Arm/Group | 100 mg CTX-4430 | 50 mg CTX-4430 | Pooled CTX-4430
Number analyzed (Participants) | 21 | 22 | 43
hazard ratio | 0.73 [0.328 to 1.641] | 0.69 [0.313 to 1.514] | 0.71 [0.359 to 1.408]

14. Other Pre Specified Outcome: Subjects Without a Pulmonary Exacerbation by Subjects if Taking CFTR-Modulator Therapy at Baseline
Description: Subjects who did not experience a protocol-defined pulmonary exacerbation during the study.
Time Frame: Week 48
Population: Population of subjects taking CFTR modulating therapy at Baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | 100 mg CTX-4430 | 50 mg CTX-4430 | Pooled CTX-4430 | Matching Placebo
Number analyzed (Participants) | 21 | 22 | 43 | 19
Participants | 10 | 10 | 20 | 6

15. Post Hoc Outcome: Number of Pulmonary Exacerbation by Baseline FEV1 Percent Predicted at Week 48
Description: as for outcome 2
Time Frame: Week 48
Population: Subject's FEV1 percent predicted at screening are presented below.
Measure: Mean (95% Confidence Interval); unit: pulmonary exacerbations per year
Arm/Group | 100 mg CTX-4430 | 50 mg CTX-4430 | Pooled CTX-4430 | Matching Placebo
Number analyzed (Participants) | 66 | 67 | 133 | 66
pulmonary exacerbations per year
  Baseline FEV1>50%: number analyzed (Participants) | 62 | 65 | 127 | 63
  Baseline FEV1>50% | 1.5094 [1.1549 to 1.9727] | 1.4376 [1.0991 to 1.8803] | 1.4731 [1.2187 to 1.7806] | 1.5297 [1.1708 to 1.9986]
  Baseline FEV1>55%: number analyzed (Participants) | 53 | 60 | 113 | 55
  Baseline FEV1>55% | 1.5006 [1.1265 to 1.9989] | 1.4159 [1.0760 to 1.8633] | 1.4576 [1.1952 to 1.7777] | 1.5425 [1.1643 to 2.0435]
  Baseline FEV1>60%: number analyzed (Participants) | 43 | 52 | 95 | 43
  Baseline FEV1>60% | 1.2698 [0.9181 to 1.7561] | 1.4446 [1.0907 to 1.9133] | 1.3544 [1.0928 to 1.6785] | 1.4728 [1.0795 to 2.0094]
  Baseline FEV1>65%: number analyzed (Participants) | 35 | 40 | 75 | 39
  Baseline FEV1>65% | 1.0473 [0.7170 to 1.5298] | 1.2523 [0.9018 to 1.7390] | 1.1452 [0.8912 to 1.4716] | 1.4489 [1.0540 to 1.9918]
  Baseline FEV1>70%: number analyzed (Participants) | 29 | 31 | 60 | 32
  Baseline FEV1>70% | 0.9198 [0.5930 to 1.4269] | 1.1995 [0.8250 to 1.7440] | 1.0504 [0.7871 to 1.4018] | 1.5365 [1.0912 to 2.1636]
  Baseline FEV1>75%: number analyzed (Participants) | 22 | 25 | 47 | 24
  Baseline FEV1>75% | 0.8417 [0.4913 to 1.4418] | 1.2786 [0.8358 to 1.9560] | 1.0374 [0.7361 to 1.4619] | 1.6125 [1.0728 to 2.4237]

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after the subject's last dose of study medication where the last dose is 48 weeks or early discontinuation of study drug.
Description: An adverse event (AE) is any untoward medical occurrence in a subject administered a pharmaceutical product and does not necessarily have a causal relationship with this product. For purposes of this trial, AEs will be reported from the signing of the study informed consent (ICF) through study completion or early termination. A Treatment-Emergent AE is an AE that occurs after the first dose of study medication.
Arm/Group | 100 mg CTX-4430 | 50 mg CTX-4430 | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/67 | 0/66
Serious Adverse Events (participants affected / at risk) | 27/66 | 26/67 | 21/66
Other Adverse Events (participants affected / at risk) | 66/66 | 67/67 | 65/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 100 mg CTX-4430 (N=66) | 50 mg CTX-4430 (N=67) | Matching Placebo (N=66)
Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Chronic Sinusitis (Infections and infestations) | 0 | 1 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 21 | 23 | 19
Lower respiratory tract infection fungal (Infections and infestations) | 1 | 0 | 0
Nocardiosis (Infections and infestations) | 0 | 0 | 1
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1
Scedosporium infection (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Borderline serous tumour of ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Antibiotic therapy (Surgical and medical procedures) | 2 | 0 | 0
Therapeutic embolisation (Surgical and medical procedures) | 0 | 0 | 1
Therapy Change (Surgical and medical procedures) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 100 mg CTX-4430 (N=66) | 50 mg CTX-4430 (N=67) | Matching Placebo (N=66)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 43 | 45 | 49
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 27 | 21
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 12 | 17 | 11
Nasopharyngitis (Infections and infestations) | 14 | 11 | 13
Headache (Nervous system disorders) | 9 | 16 | 7
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 7 | 13 | 11
Fatigue (General disorders) | 9 | 9 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 7 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | 9
Pyrexia (General disorders) | 8 | 6 | 7
Diarrhoea (Gastrointestinal disorders) | 5 | 9 | 4
Nausea (Gastrointestinal disorders) | 8 | 5 | 5
Chest discomfort (General disorders) | 8 | 3 | 7
Abdominal pain upper (Gastrointestinal disorders) | 3 | 7 | 5
Sinusitis (Infections and infestations) | 6 | 3 | 5
Vomiting (Gastrointestinal disorders) | 3 | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 4
Constipation (Gastrointestinal disorders) | 1 | 4 | 3
Gastroenteritis (Infections and infestations) | 4 | 1 | 2
Influenza (Infections and infestations) | 5 | 3 | 4
Rhinitis (Infections and infestations) | 3 | 4 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 4 | 5
Alanine aminotransferase increased (Investigations) | 4 | 0 | 2
Forced expiratory volume decreased (Investigations) | 5 | 4 | 4
Sputum Abnormal (Investigations) | 0 | 4 | 1
Weight decreased (Investigations) | 1 | 4 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 5
Rash (Skin and subcutaneous tissue disorders) | 6 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication or (2) 24 months after close of the study, whichever occurs first.

Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 90 days (which may be extended under certain circumstances related to protection of intellectual property as well as for deletion of any Confidential Information).

DOCUMENTS (2):
  • Study Protocol (2016-05-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT02443688/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT02443688/SAP_001.pdf